CLINICAL TRIAL: NCT03642834
Title: A Phase I, Open-Label Study to Assess the Safety, Tolerability, Pharmacokinetics of ICP-105 in Patients With Advanced Solid Malignancies
Brief Title: Study of ICP-105 in Solid Tumors Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00201
Record Dates: First submitted 2018-08-17; First posted 2018-08-22 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP-105 Single Arm (Experimental): ICP-105 of multiple dose levels, dose escalation steps may be modified based on the safety from the previous dose.
  Interventions: Drug: ICP-105

INTERVENTIONS:
Drug: ICP-105 — 25mg, 100mg capsule

SUMMARY:
Open-label, non-randomized, Phase I, dose-escalating, first-in-man study.

DETAILED DESCRIPTION:
The study consisted of a screening period, a treatment period with repeated 28-day treatment cycles (duration treatment with ICP-105), and a follow-up period (within 30 days of the last dose and post-treatment follow-up 30 days after the last visit). The recruited patients receive a single dose on day 1, then after a 3-day washout period, multiple dosing will be initiated following dose-escalation schedule. The dose-limiting toxicity (DLT) assessment period consisted of Cycle 0 (single dose and washout period) and Cycle 1 (28-day cycle).

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
* At least one evaluable disease according to RECIST1.1.
* Histologically or cytologically confirmed solid tumors, failure to respond to standard therapy, or for whom standard therapy does not exist.
* Adequate bone marrow, liver, renal, and cardiovascular function.

Exclusion Criteria:

* Previous treatment with FGF19, FGFR4 inhibitors and/or pan-FGFR inhibitors.
* Anti-cancer therapy, such as chemotherapy, immunotherapy, hormonal, targeted therapy, or investigational agents within four weeks of the first dose of ICP-105.
* Major surgery within 6 weeks of the first dose of ICP-105.
* Significant GI disorder(s) that could interfere with the absorption, metabolism, or excretion of ICP-105.
* Crohn's disease with symptoms and systemic treatment.
* Central nervous system (CNS) metastasis.
* Current clinically significant cardiovascular disease including:
* Any class 3 or 4 cardiac disease such as arrhythmia, congestive heart failure or myocardial infarction defined by the New York Heart Association Functional Classification, or left ventricular ejection fraction (LVEF) < 50%, Primary cardiomyopathy, clinical significant QTc prolong history or QTc>470ms (female) QTc>450ms (male).
* Known active bleeding within 2 months of screening or 6 months of bleeding history.
* Lung function impairment by pleural effusion or ascites, any history of interstitial pneumonia, deep vein thrombosis, pulmonary embolism.
* Known active infection with HBV, HCV or HIV or any uncontrolled active systemic infection.
* Non-hematological toxicity must recover to ≤ Grade 1 from prior anti-cancer therapy (excluding alopecia, nausea and vomiting).
* Lactating or pregnant women, or women who will not use contraception during the study and for 180 days after the last dose of study drug if sexually active and able to bear children.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Every cycle (28 days) for approximately 24 months or earlier if patient terminates from the study
  will be evaluated by CTCAE v4.03

SECONDARY OUTCOMES:
Cmax | Every cycle (28 days) for approximately 24 months or earlier if patient terminates from the study
  the peak plasma concentration
AUC | Every cycle (28 days) for approximately 24 months or earlier if patient terminates from the study
  area under the plasma concentration vs. time curve
Apparent half-life for designated elimination phases (t½) | Every cycle (28 days) for approximately 24 months or earlier if patient terminates from the study
  will be measured and calculated with noncompartmental analysis using WinNonlin

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, PhD, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China